CLINICAL TRIAL: NCT07063134
Title: Investigation of the Relationship Between Chronic Mouth Breathing and SARS-CoV-2 Positivity in the Pediatric Population
Brief Title: Chronic Mouth Breathing and SARS-CoV-2 Positivity in the Pediatric Population
Acronym: BREATH-COV
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Serap Titiz Yurdakal, Associate Professor of Orthodontics, Dokuz Eylul University
Other Study IDs: DEUORTO-CMB-2025
Record Dates: First submitted 2025-06-26; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: SARS-CoV-2 Infection
Keywords: Coronavirus- Mouth breathing - Nasal breathing - Delta variant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Positive Group: Participants who tested positive for SARS-CoV-2 by PCR at the time of evaluation.
- COVID-19 Negative Group: Participants who tested negative for SARS-CoV-2 by PCR at the time of evaluation.

SUMMARY:
Numerous non-scientific articles on the internet assert the significance of nasal breathing in protecting against COVID-19. Although nasal breathing is anticipated to result in a reduced intake of bioparticles when compared to mouth breathing due to the filtering mechanisms present in the nasal cavity, we have yet to identify any in vivo studies within the literature that definitively ascertain the correlation between mouth breathing and COVID-19 positivity. Consequently, this study aimed to investigate the impact of chronic mouth breathing on testing positive for COVID-19 in children.

DETAILED DESCRIPTION:
Objective Coronavirus disease (COVID-19) is an infectious respiratory illness caused by the SARS-CoV-2 virus. Breathing patterns may influence the transmission of respiratory diseases. Mouth breathing inhaled pollutants and pathogens directly into the lungs. Therefore, this research investigated the impact of chronic mouth breathing on COVID-19 positivity in children.

Materials and Methods A total of 173 patients aged between 10 and 17 years, without any systemic diseases or COVID-19 vaccinations, who were undergoing COVID-19 testing, were included in the study. The age, gender, simplified oral hygiene index, and respiratory models of the included patients were assessed. Patients with a specific malocclusion caused by mouth breathing were diagnosed as "mouth breathers" through clinical assessments. Those who tested positive for COVID-19 were assigned to the experimental group, while those who tested negative were designated as the control group. The differences in mouth breathing rates, simplified oral hygiene index, and sociodemographic data (sex and age) between groups were statistically analysed. Subsequently, the relationship between mouth breathing and the Delta variant was examined.

Results No statistically significant differences were found in sex, breathing pattern, and the simplified oral hygiene index, except for age (p>0.05). The average age of the patients in the experimental group was lower. The Delta variant was more common among chronic mouth breathers (p<0.05).

Conclusion Chronic mouth breathing heightens the risk of transmission, as the pathogenicity of COVID-19 viruses increases.

Clinical relevance Healthcare professionals should possess the knowledge necessary to identify individuals who breathe through their mouths, as this group faces a heightened risk of contracting respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* tested for COVID-19

Exclusion Criteria:

* Not tested for COVID-19

Ages: 10 Hours to 18 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 173 patients aged between 10 and 17 years, without any systemic diseases or COVID-19 vaccinations, who were undergoing COVID-19 testing, were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Rate of COVID-19 Positivity in Chronic Mouth Breathers Compared to Nasal Breathers | At 2 weeks post-COVID-19 recovery"
  Proportion of COVID-19 positivity among chronic mouth breathers compared to nasal breathers

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University Faculty of Dentistry, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided